CLINICAL TRIAL: NCT02068521
Title: An Open-Label, Long-Term Safety Study of A Long-acting Human Growth Hormone Somavaratan (VRS-317) in Children With Growth Hormone Deficiency
Brief Title: Versartis Long-Term Safety Study of Somavaratan
Acronym: VISTA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The primary endpoint of non-inferiority to daily therapy in the pediatric Phase 3 study was not achieved
Sponsor: Versartis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13VR3
Record Dates: First submitted 2014-02-06; First posted 2014-02-21 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Pediatric Growth Hormone Deficiency
Keywords: Growth Hormone Deficiency; Pediatric Growth Hormone Deficiency; GHD; PGHD; VRS-317; Versartis; Growth disorder; Long acting growth hormone; Growth hormone; Weekly growth hormone dosing; Semi-monthly growth hormone dosing; Monthly growth hormone dosing; IGF-I; Short stature; Height velocity; Annual height velocity; Growth rate; Somavaratan
MeSH Terms: conditions — Dwarfism, Pituitary; Growth Disorders; Dwarfism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment naive subjects with GHD (Experimental): Up to 100 new treatment naïve subjects with GHD will receive somavaratan 3.5mg/kg twice monthly.
  Interventions: Drug: somavaratan
- Subjects who have completed a somavaratan study (Experimental): All subjects after participation in (12VR2) or participation in the 14VR4 protocols have the option to receive somavaratan 3.5mg/kg twice monthly.
  Interventions: Drug: somavaratan

INTERVENTIONS:
Drug: somavaratan — Subcutaneous injection
  Other Names: VRS-317

SUMMARY:
Protocol 13VR3 is is a multi-center, open-label study assessing long-term somavaratan administration.

Patients will be monitored for safety throughout their participation in the study. Safety will be monitored by physical examination, inspection of injection sites, vital signs, clinical laboratory determinations (including fasting glucose, insulin, and lipids), 12-lead ECGs (for new treatment naïve subjects and subjects not previously exposed to somavaratan), PK/PD assessments, and immunogenicity assessments.

Adverse events (AEs) and concomitant medications will be captured. AEs will be coded using CTCAE v 4.0. AEs will be coded using the MedDRA dictionary and CMs using the WHO Drug dictionary.

DETAILED DESCRIPTION:
Protocol 13VR3 is a multi-center, open-label study assessing long-term somavaratan administration. It is open to subjects completing a somavaratan study in children with growth hormone deficiency (GHD), as well as up to 100 new treatment naïve subjects with GHD. All subjects will receive somavaratan 3.5 mg/kg twice monthly. The study will be conducted at approximately 70 Pediatric Endocrinology centers in the United States, Canada, and Europe.

ELIGIBILITY:
Inclusion Criteria for Subjects Completing a Previous Somavaratan Study:

1. Completion of a somavaratan clinical study.
2. Willing and able to comply with all study procedures.

Exclusion Criteria for Subjects Completing a Previous somavaratan Study:

1. Withdrawal from a somavaratan clinical study.
2. Use of certain medications with potential to alter responses to the test product.
3. Presence of a significant medical condition.

Inclusion Criteria for New Treatment Naïve Subjects:

1. Chronological Age ≥ 3.0 years.
2. Pre-pubertal status.
3. Diagnosis of GHD as documented by two or more GH stimulation test results ≤ 10.0 ng/mL.
4. Normal thyroid function at Screening Visit in subjects not being treated for hypothyroidism.
5. Normal adrenal function at Screening Visit or within 6 months of the Screening Visit, in subjects not being treated for adrenal insufficiency. Subjects with adrenal insufficiency must receive glucocorticoid treatment for a minimum of 4 weeks before study drug administration.
6. Pathology relating to cause of GHD must be stable for at least 6 months prior to screening.
7. Legally authorized representatives must be willing and able to give informed consent.

Exclusion Criteria for New Treatment Naïve Subjects:

1. Prior/concomitant treatment with any growth promoting agent.
2. Current, significant disease.
3. Chromosomal aneuploidy, significant gene mutations or confirmed diagnosis of a named syndrome.
4. Birth weight and/or birth length less than 5th percentile for gestational age.
5. Prolonged daily use of anti-inflammatory doses of oral glucocorticoids.
6. Prior history of malignancy.
7. Treatment with an investigational drug in the 30 days prior to screening.
8. Known allergy to constituents of the study drug formulation.
9. Ocular findings suggestive of increased intracranial pressure and/or retinopathy at screening.
10. Significant spinal abnormalities including scoliosis, kyphosis, Chiari malformation, and spina bifida variants.
11. Significant abnormality in screening studies.
12. History of pancreatitis or undiagnosed chronic abdominal pain.
13. History of spinal or total body irradiation.
14. Other pituitary hormone deficiencies that are not properly treated.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 4 years
  Safety assessments include recording of adverse events and concomitant medications, monitoring of injection sites, vital signs and clinical laboratory determinations.

OTHER OUTCOMES:
Evaluate the changes in pharmacodynamics (PD) responses, bone age, weight, height velocity, height standard deviation scores, metabolic parameters, pubertal development and anti-drug antibody responses during long-term somavaratan treatment | Up to 4 years
  PK/PD peak and trough measurements will be assessed throughout the study with assessment of plasma VRS-317 concentrations and IGF-I and its binding proteins measured at pre-specified time points.

CONTACTS AND LOCATIONS:
Overall Officials: Will Charlton, MD, Study Director — Versartis Inc.

REFERENCES:
- See also: Versartis website — http://versartis.com